CLINICAL TRIAL: NCT03753035
Title: Observance of Anticonvulsant Treatments and Quality of Life of Epileptic Children
Acronym: ObEPI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: ObEPI
Record Dates: First submitted 2018-11-22; First posted 2018-11-26 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Epilepsy; Children, Only; Quality of Life; Seizures; Patient Compliance
Keywords: epilepsy; children; seizures; patient compliance; quality of life
MeSH Terms: conditions — Epilepsy; Seizures; Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- epileptic children: Completion of questionnaire, during medical consultation, on compliance and quality of life

SUMMARY:
There is little epidemiological data in the literature on the therapeutic compliance of epileptic children. Yet it is a fundamental issue in the therapeutic education and balance of this pathology. To obtain more epidemiological precision on the observance of epileptic children and to propose, according to the factors involved, the improvement of practices (therapeutic education ..). Propose an evaluation of the quality of life of their children by a suitable self-questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* • Child aged 5 to 17

  * Child who has received complete information on the organization of the research and who has not objected to his participation and the exploitation of his data
  * Holder (s) of the parental authority present (s) having received the complete information on the organization of the research and not being opposed to the participation and the exploitation of the data of his child
  * Epileptic child
  * Follow-up at the neuro pediatric department of CHRU Nancy

Exclusion Criteria:

* epileptic encephalopathy
* Multiply handicapped child

Ages: 5 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: all epileptic children at Nancy Children Hospital
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2018-11-29 (Actual); Primary Completion 2019-04-30 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
Mean compliance | 6 months
  Mean compliance score measured by the validated Modified Morisky Medication Adherence Scales 8 for epileptic patients 11 subscale with a 5-point Likert scale. According to the scoring system for the MMAS, 8=high adherence, 6 to <8=medium adherence, and <6=low adherence. Patients who had a low or a moderate rate of adherence were considered nonadherent5.

SECONDARY OUTCOMES:
Compliance score of the modified Modified Morisky Medication Adherence Scales 8 | 6 months
  distribution of responses to new items of the modified MMAS8 scale, internal structure)
quality of life of epileptic children | 6 months
  Quality of life score measured by the IImpact of Pediatric Epilepsy Scale An 11-item scale was created for children and/or parents' use (according to age) to evaluate the influence of epilepsy on the major aspects of their family and child's life 5 items scale with a 5 point Likert scale
syndromes | 6 months
  MMAS8 compliance score according to syndromes and equilibrium of epilepsy

CONTACTS AND LOCATIONS:
Locations (1):
- GIRARD, Nancy, Lorraine, France